CLINICAL TRIAL: NCT05052281
Title: Promoting Healthy Brain Development Via Prenatal Stress Reduction: An Innovative Precision Medicine Approach
Brief Title: Promoting Healthy Brain Development: Wellness for 2 Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: Ann & Robert H Lurie Children's Hospital of Chicago (Other)
Responsible Party: Principal Investigator, Lauren Wakschlag, PhD, Professor, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB 2019-2515
Record Dates: First submitted 2019-08-30; First posted 2021-09-22 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Prenatal Stress
Keywords: Pregnancy; Pre-natal; Post-Natal; Neurodevelopment

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Intervention group (Experimental): The first MB course session and technology training will take place in-person, prior to 23 weeks gestation. The Mothers and Babies course (MB) is a 12-session manualized stress-reduction intervention that will be delivered to participants, prenatally, with an integrated technology suite designed for timely detection and response to maternal stress. Sessions are delivered 1-on-1 with a trained facilitator and are based on principles of cognitive-behavioral therapy (CBT) and attachment theory. The MB course is divided into 3 sections: 1) Pleasant Activities; 2) Thoughts; 3) Contact with Others. Throughout each module, mindfulness skills training will be integrated as a strategy to help "center" participants. All participants will receive a Participant Manual for Families, containing worksheets that correspond to the 12 sessions.
  Interventions: Behavioral: Mothers and Babies (MB) Course; Behavioral: Just in Time Intervention (JITI) Content; Device: Biostamp nPoint Device
- Stress monitoring (control) group (Active Comparator): This group will not receive any additional intervention but will engage in stress monitoring via biosensors and EMA text messages through the 14 week period
  Interventions: Device: Biostamp nPoint Device

INTERVENTIONS:
Behavioral: Mothers and Babies (MB) Course — The Mothers and Babies course (MB) is a 12-session manualized stress-reduction intervention that will be delivered to participants, prenatally, with an integrated technology suite designed for timely detection and response to maternal stress.
  Arms: Intervention group
Behavioral: Just in Time Intervention (JITI) Content — Participants will also receive additional MB intervention content in the form of "just-in-time" text messages, which will be sent to participants' smartphones every other day for up to 12 weeks. During the current trial, participants will receive text message prompts with links to additional stress reduction content based on a combination of their objective (sensor) and subjective (EMA) stress responses from the previous day.
  Arms: Intervention group
Device: Biostamp nPoint Device — During the intervention period, participants will be asked to wear the BioStamp nPoint sensor, daily, while engaging in their usual activities (e.g., sleep, showering, exercise). The BioStamp Sensor is a thin, wearable patch, equipped with wireless high-range 6-axis gyroscope + accelerometer, and sEMG and ECG sensors, that adheres to the skin using a disposable medical-grade adhesive sticker (with adhesive similar to Band-Aid).

SUMMARY:
The "Promoting Healthy Brain Project" (PHBP) is part of the Lurie Children's Hospital Strategic Research Initiative on Perinatal Origins of Childhood Disease: Research & Prevention at the Maternal-Fetal Interface. The overall purpose of the PHBP is to test whether reducing maternal stress during pregnancy is associated with improved neurodevelopment in the first year of life. This will be tested via a randomized controlled trial (n = 100) of a technology and mindfulness enhanced prenatal stress-reduction intervention (Mothers and Babies; MB).

DETAILED DESCRIPTION:
The "Promoting Healthy Brain Project" (PHBP) aims to improve infant neurodevelopmental trajectories by intervening on the fetal environment. The PHBP will experimentally test whether reducing prenatal maternal stress is associated with improved neurodevelopment in the first year of life. A randomized controlled trial (RCT) of a technology and mindfulness-enhanced prenatal maternal stress-reduction intervention (The Mothers and Babies Course; MB), compared to usual prenatal care. Prospective evaluation of infant neurodevelopmental outcomes will take place through infant age 24 months. Participants assigned to the intervention group will be offered the 12-session MB intervention, a well-studied intervention that will include new mindfulness practice enhancements designed to promote practice of awareness and attention to the present moment. MB visits will be delivered 1-on-1 by a trained facilitator in an open and nonjudgmental way, and will be offered in-person, over the phone, and/or by video chat. Throughout the intervention, all participants (intervention group and control group) will also wear a wireless, "smart" health sensing device (BioStamp Sensor - nPoint Device) that will measure heart rate and motion. Mothers' heart rate variability and self-reported stress and emotion will be monitored using the BioStamp Sensor and brief smartphone surveys. For mothers in the intervention group, patterns of prolonged stress will trigger a "just-in-time adapted intervention" (JITAI) that will be delivered to mothers' smartphones. The booster intervention will include activities that will enhance skills learned in the MB course. All participants will complete self-report measures of prenatal maternal stress, emotion, depression, and skills related to the intervention (e.g., mindfulness). Infant neurodevelopmental health will be measured via brain and behavioral indicators of self-regulation, including performance-based indicators of executive function and corollary prefrontal cortex maturation and dimensional phenotypes of disruptive behavior, particularly irritability.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years old;
* enrolled under 22 weeks gestation;
* receiving prenatal care from a Northwestern University prenatal care clinic & planning to deliver at Northwestern Hospitals;
* English-speaking
* Participants must own a smartphone and be must be willing to receive text messages and respond to short online surveys using their smartphone.
* Eligible participants must also agree to wear a wireless adhesive sensor, the BioStamp, daily, throughout the 12-week MB course.
* Eligible participants will also have WiFi internet access for the duration of their participation in the study, in order to complete online questionnaires and upload sensor data.
* Eligible participants must also agree to have their child participate in the neurodevelopmental assessments from birth-12 months.

Exclusion Criteria:

* Women will be ineligible to participate in this study if they have known pregnancy or chronic medical complications that may place their infant at risk for neurological disorders (e.g., HIV; acute cytomegalovirus infection (CMV); toxoplasmosis; zika virus; Phenylketonuria (PKU); chromosomal anomalies; metabolic disorder; substance use disorders) or significant mental health disorders (e.g., schizophrenia, bipolar disorder, psychosis) which could interfere with study adherence.
* Participants unable to wear the BioStamp Sensor due to known skin sensitivity (e.g., allergy to adhesives or silicone), current skin irritation, or broken skin at the placement site will not be eligible to participate.
* Participants with a pacemaker or other sensitive medical device will be excluded.
* Women will not be eligible to participate if unable to provide informed consent, complete MB sessions, or complete study assessments in English.
* Women who are currently participating in an MB course at the time of recruitment will not be eligible to participate.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2019-07-15 (Actual); Primary Completion 2024-07-28 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
Disruptive Behavior Diagnostic Observation Schedule (DB DOS) | 12 months, 24 months
  The DB DOS is a standardized observation of infant arousal, soothability, reactivity, and temper loss. During early infancy, the
Perceived Stress Scale (PSS) | Prenatal, 1 month, 3 months, 7 months, 12 months, 24 months
  The PSS is a self-report measure of the degree to which an individual perceives their life situations to be stressful. The instrument includes 10 items that assess how unpredictable, uncontrollable, and overloaded respondents find their lives, and assess current levels of experienced stress.
MAP-DB | 1 month, 7 months, 12 months, 24 months
  Parent report measure of infant irritability.
PROMIS Depression | Prenatal, 1 month, 3 months, 7 months, 12 months, 24 months
  Mothers complete a 28-item scale that assesses depressive symptoms experienced in the past 7 days.
State Trait Anxiety Inventory (STAI) | Prenatal, 1 month, 3 months, 7 months, 12 months, 24 months
  The STAI is a 40 item self report questionnaire that assesses both state anxiety and trait anxiety.

SECONDARY OUTCOMES:
Five Facet Mindfulness Questionnaire (FFMQ) | Prenatal, 1 month, 3 months, 7 months, 12 months, 24 months
  The FFMQ is a 39-item self report survey that taps into five areas of mindfulness, including observation, description, aware actions, non-judgmental inner experience, and non-reactivity.
NICU Neonatal Behavioral Scale (NNNS) | 1 month
  The NNNS is an assessment of neurobehavioral organization, neurological reflexes, motor development - active and passive tone, and signs of stress and withdrawal in neonates, developed for use with at-risk or drug-exposed infants but has been normed with typically developing infants.
Test of Infant Motor Performance (TIMP) | 1 month
  The TIMP is a norm-referenced measure designed to evaluate motor control and organization of posture and movement for functional activities in infants 32 weeks gestational age to four months post-term age and measures both spontaneous behaviors and elicited items.
General Movements Assessment (GMA) | 1 month
  General movements are a developmentally regulated pattern of spontaneous motor activity. By 10-15 weeks of age, the predominant general movements seen are called Fidgety Movements - a pattern of continuous, small amplitude movements of the neck, trunk and limbs during wakefulness that disappear with agitation. These patterns are identifiable and are classified as normal if present (intermittent or continual), and abnormal if exaggerated (with respect to speed and amplitude), sporadic (interspersed with long pauses) or absent. Babies are observed for up to 30 minutes in a supine position to assess for spontaneous movements.
Alberta Infant Motor Scale (AIMS) | 1 month
  The Alberta Infant Motor Scale (AIMS) is a 10-20 minute norm referenced, standardized, gross motor assessment. Infants are observed in four positions: prone, sitting, supine, and standing. For each subscale, items are scored as "observed" or "not observed". A total raw score and percentile are calculated.
Maternal Heart Rate Variability | Pregnancy (duration 14 weeks)
  variability/physiological stress as indicated by a machine learned model applied to electrocardiogram (ECG) signals.
Prefrontal cortex thickness | 1 month, 12 months, 24 months
  Cortical thickness and surface area of pre-frontal cortex regions, which have been linked to child irritability and Infant dysregulation, is measured through natural sleep MRI.
Inflammatory and neuroimmune biomarkers | At birth
  Placenta and cord blood will be collected at birth. Tests to be performed on these samples include measurement of inflammatory markers related to stress, such as a multiplex immunoassay panel of the following cytokines and chemokines: (IL-6, IL-8, IL-10, C-reactive protein, TNF-alpha, TGF-beta, IL-1beta, procalcitonin, cortisol).
EEG power | 1 month, 12 months, 24 months
  The baby will complete a baseline or resting EEG for 2-5 minutes and then hear an auditory oddball paradigm with speech syllables while resting for ~10 min. EEG (electroencephalogram) power will be measured as a marker infant neurodevelopment.
ERP mean amplitude | 1 month, 12 months, 24 months
  The baby will complete a baseline or resting EEG for 2-5 minutes and then hear an auditory oddball paradigm with speech syllables while resting for ~10 min. ERP (event related potential) mean amplitude will be measured as a marker of infant neurodevelopment.
Birthweight | Birth
  Infant birthweight will be obtained from EHR data collected at the hospital at birth
Maternal Infant Responsiveness Instrument (MIRI) | 1 month, 7 months, 12 months
  The MIRI is a 22 item questionnaire designed to assess a mother's feelings about her infant, her recognition of her responsiveness to the infant, and her infants responses.
Infant Behavior Questionnaire-Revised (IBQ-R) short form | 1 month, 7 months, 12 months
  The IBQ-R is a parent-report survey designed to measure multiple dimensions of temperament in infants up to age 12 months.
Bayley Scales of Infant Development | 7 months, 12 months, 24 months
  The Bayley Scales of Infant and Toddler Development Fourth Edition (Bayley-4) is a five-domain assessment tool used to determine developmental delays in children. The developmental domains are cognitive, language, motor, social-emotional, and adaptive behavior, and include direct assessment of the child and parent report.
Preschool Age Psychiatric Assessment (PAPA) | 24 months
  Parent structured interview for diagnosing psychiatric disorders in children ages 2-5.
Brief Infant Toddler Social Emotional Assessment (BITSEA) | 12 months, 24 months
  Parent report measure of behavior problems and social competencies in children ages 1-3 that identifies delays or deficits in areas of social-emotional development.
Early Childhood Irritability Related Impairment Interview (E-CRI) | 24 months
  The E-CRI is a semi-structured interview designed to measure early childhood impairment resulting from young children's tantrums and irritability across various contexts.
Perceived Stress Scale (PSS) | 1 month, 3 months, 7 months, 12 months, 24 months
  Self-report measure of the degree to which an individual perceives their life situations to be stressful. The instrument includes 10 items that assess how unpredictable, uncontrollable, and overloaded respondents find their lives, and assess current levels of experienced stress.
Behavioral Activation Depression Scale (BADS) - short form | prenatal, 3 months, 7 months, 12 months, 24 months
  Self-report 9-item measure of behaviors that indicate depression and can be targeted for change by cognitive behavioral therapy and behavior activation. Mothers complete this measure regarding behaviors experienced over the past week.
Negative Mood Regulation Scale (NMRS) | prenatal, 3 months, 7 months, 12 months, 24 months
  This self-report, 30-item scale measures expectancies and beliefs that the mothers have regarding their abilities to alleviate their negative mood, anger, anxiety and depression.
Parenting Stress Index (PSI) - Role Restriction Subscale | 3 months, 7 months, 12 months, 24 months
  The PSI Role Restriction subscale includes 7 mother-report items regarding her feelings of limited freedom and restriction of her identity to the parenting role.
Parental Cognitions and Conduct Toward the Infant Scale (PACOTIS) | 1 month, 3 months, 7 months, and 12 months
  The PACOTIS is a mother report measure of their actions, thoughts, and feelings during interactions with their baby.
MacArthur-Bates Communicative Development Inventories (MCDI) | 12 months, 24 months
  The MCDI is a parent-report questionnaire about their child's communication and language development. The Words & Gestures form is used at 12 months and the Words & Sentences form is used at 24 months.
Medical Outcomes Study (MOS) Social Support Survey | Prenatal, 3 months, 7 months, 12 months, 24 months
  The MOS Social Support Survey is a 19-item self-report measure of the mother's availability of social support in a variety of domains including emotional support, tangible support, affectionate support, and positive social interaction.

OTHER OUTCOMES:
Family Life Impairment Scale (FLIS) | 12 months, 24 months
  The FLIS is a parent report survey that assesses the degree to which a child's behavior impacts the family's ability to participate in typical activities.
PROMIS Anxiety | Prenatal, 1 month, 3 months, 7 months, 12 months, 24 months
  Mothers complete the PROMIS Anxiety scale, which includes items that assess fear, anxious misery, hyperarousal, and somatic symptoms related to anxiety.
Family Relationship Index (FRI) | prenatal, 3 months, 7 months, 12 months, 24 months
  The FRI is a 12-item survey designed to assess family cohesion, communication and conflict-resolution.

CONTACTS AND LOCATIONS:
Overall Officials: Lauren Wakschlag, PhD, Principal Investigator — Northwestern University
Locations (2):
- United States (2):
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Northwestern University (Feinberg School of Medicine), Chicago, Illinois

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be shared with other investigators. Investigators from outside the study will be asked to sign an agreement of confidentiality in order to receive the data requested. Data will be stored for at least 7 years. We plan to archive the de-identified data in a data repository for future use by other researchers, after the study is completed. Additionally, data from this study will be used in the Mental Health Earlier Synthetic Cohort (MHESC) Study in order to generate a pragmatic clinical risk calculator to predict preschool psychopathology. MHESC pools three extramural cohorts at Northwestern University and Washington University in St. Louis, one of which is the Wellness for 2 Study to form a clinically enriched "synthetic" cohort. Therefore, data will be shared with authorized individuals at Washington University.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be stored for at least 7 years.

REFERENCES:
- [Background] Talge NM, Neal C, Glover V; Early Stress, Translational Research and Prevention Science Network: Fetal and Neonatal Experience on Child and Adolescent Mental Health. Antenatal maternal stress and long-term effects on child neurodevelopment: how and why? J Child Psychol Psychiatry. 2007 Mar-Apr;48(3-4):245-61. doi: 10.1111/j.1469-7610.2006.01714.x. PMID 17355398
- [Background] Kinsella MT, Monk C. Impact of maternal stress, depression and anxiety on fetal neurobehavioral development. Clin Obstet Gynecol. 2009 Sep;52(3):425-40. doi: 10.1097/GRF.0b013e3181b52df1. PMID 19661759
- [Background] O'Connor TG, Heron J, Golding J, Glover V; ALSPAC Study Team. Maternal antenatal anxiety and behavioural/emotional problems in children: a test of a programming hypothesis. J Child Psychol Psychiatry. 2003 Oct;44(7):1025-36. doi: 10.1111/1469-7610.00187. PMID 14531585
- [Background] de Bruijn AT, van Bakel HJ, van Baar AL. Sex differences in the relation between prenatal maternal emotional complaints and child outcome. Early Hum Dev. 2009 May;85(5):319-24. doi: 10.1016/j.earlhumdev.2008.12.009. Epub 2009 Jan 21. PMID 19162414
- [Background] Grizenko N, Fortier ME, Zadorozny C, Thakur G, Schmitz N, Duval R, Joober R. Maternal Stress during Pregnancy, ADHD Symptomatology in Children and Genotype: Gene-Environment Interaction. J Can Acad Child Adolesc Psychiatry. 2012 Feb;21(1):9-15. PMID 22299010
- [Background] Mendelson T, Leis JA, Perry DF, Stuart EA, Tandon SD. Impact of a preventive intervention for perinatal depression on mood regulation, social support, and coping. Arch Womens Ment Health. 2013 Jun;16(3):211-8. doi: 10.1007/s00737-013-0332-4. Epub 2013 Mar 2. PMID 23456540
- [Background] Tandon SD, Leis JA, Mendelson T, Perry DF, Kemp K. Six-month outcomes from a randomized controlled trial to prevent perinatal depression in low-income home visiting clients. Matern Child Health J. 2014 May;18(4):873-81. doi: 10.1007/s10995-013-1313-y. PMID 23793487
- [Background] Tandon SD, Perry DF, Mendelson T, Kemp K, Leis JA. Preventing perinatal depression in low-income home visiting clients: a randomized controlled trial. J Consult Clin Psychol. 2011 Oct;79(5):707-12. doi: 10.1037/a0024895. PMID 21806298
- [Derived] Tandon SD, Moskowitz JT, Edwards RC, Zhang Y, Giase G, Sinche B, Blum AL, Krislov S, Reynolds HM, Rangarajan A, Cummings P, Petitclerc A, Alshurafa N, Grobman WA, Ward EA, Wakschlag LS. Effects of a Personalized Stress Management Intervention on Maternal Mental Health: A Randomized Clinical Trial. Arch Womens Ment Health. 2025 Dec;28(6):1585-1595. doi: 10.1007/s00737-025-01619-5. Epub 2025 Sep 17. PMID 40960524